CLINICAL TRIAL: NCT04236622
Title: Clinical and Radiographic Evaluation of Dental Implants Installed Between 2004 and 2010
Acronym: implants
Status: Completed | Type: Observational
Sponsor: Universidade Metropolitana de Santos (Other)
Responsible Party: Principal Investigator, CAIO VINICIUS G. ROMAN TORRES, Professor, Universidade Metropolitana de Santos
Other Study IDs: SantosMU6
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Dental Implant Failed
Keywords: dental implants; periodontal index; peri-implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health: For each patient we evaluated the Probing Depth (PD), measured in mm, and the following dichotomous variables: plaque index (absent or present), gingival index (absent or present), occurrence of annual maintenance (absent or present), tooth position (anterior or posterior) and the patient's smoking habit (absent or present).
  Interventions: Other: Periodontal clinical exam
- Peri-implantitis: For each patient we evaluated the Probing Depth (PD), measured in mm, and the following dichotomous variables: plaque index (absent or present), gingival index (absent or present), occurrence of annual maintenance (absent or present), tooth position (anterior or posterior) and the patient's smoking habit (absent or present).
  Interventions: Other: Periodontal clinical exam

INTERVENTIONS:
Other: Periodontal clinical exam — The individuals will be submitted to a complete periodontal examination, with measurements obtained at four points per tooth and dental implant (mesial, distal, buccal and lingual / palatal), in all teeth / implants present, except for the third molars, the parameters evaluated will be: Probing Depth, Clinical Insertion Level, Plaque Index, Teeth Bleeding Index. The implants will be evaluated according to the parameters: presence of suppuration, probing depth, bleeding to probing and presence of biofilm around the implants. To perform the clinical examinations, the following instruments will be required: Willians millimeter probe, exploratory probe and clinical mirror.
  In all participants, complete periapical radiographic examinations with 14 radiographs will be performed to verify the bone cortical height level and to assist in the periodontal diagnosis.
  Other Names: Radiographic exam

SUMMARY:
The convenience sample to be included in the present study will consist of all individuals who had implants installed at the Dentistry Clinic of the University Santo Amaro, between the years 2004 and 2010. The following criteria will be evaluated: age; sex; presence of systemic disease; area in which the implant was installed; implant diameter and height; type of prosthesis installed; presence of bone resorption and annual maintenance.

DETAILED DESCRIPTION:
The control of biofilm around implants is fundamental to the success of implant therapy, and it is the duty of the dentist to inform, guide and maintain patients in order to avoid pathological processes that may lead to the loss of the implanted component. The objective of the present study will be to evaluate by clinical and radiographic parameters the condition of oral implants placed for more than five years. The convenience sample to be included in this study will be composed of all individuals who had implants installed at the Dental Clinic of the University Santo Amaro, between 2004 and 2010. The following criteria will be evaluated: age; sex; presence of systemic disease; area in which the implant was installed; implant diameter and height; type of prosthesis installed; presence of bone resorption and annual maintenance. The success and survival rate of implants through the following parameters: pain; mobility; card index (IP); bleeding rate (IS); probing depth (PS); probing bleeding (SS) that will be measured on four faces by implant: mesial, buccal, distal and lingual / palatine. For the evaluation of bone loss, a conventional periapical radiograph will be performed at the moment of patient recall. Radiographs will be scanned and analyzed using Image Tool software to verify and determine the resulting linear distance between the implant shoulder and the bone crest. Factors such as smoking, annual maintenance appointments will be related to the presence of peri-implantitis.

ELIGIBILITY:
Inclusion Criteria:

* After evaluation, individuals may be allocated into groups according to the characteristics observed, for example: carriers of single implants, patients with overdentures, individuals with systemic diseases, smokers.

Exclusion Criteria:

* Individuals who need to use or suspend systemic medication to perform the proposed clinical exams will be excluded from the study.

Ages: 30 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals of both genders, between 30 and 70 years of age, with implants placed from 2004 to 2010 will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-02-10 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Probing depth | 10 years
  lower probing depth in patients who underwent annual maintenance

SECONDARY OUTCOMES:
Plaque control | 10 years
  lower plaque index in patients who underwent annual maintenance

CONTACTS AND LOCATIONS:
Overall Officials: CAIO VINICIUS G ROMAN TORRES, PhD, Principal Investigator — University of South Australia
Locations (1):
- University of Santo Amaro - UNISA/SP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared with other researchers. The study participants allowed the use of data only for this study and for this researcher

REFERENCES:
- [Result] van Velzen FJ, Ofec R, Schulten EA, Ten Bruggenkate CM. 10-year survival rate and the incidence of peri-implant disease of 374 titanium dental implants with a SLA surface: a prospective cohort study in 177 fully and partially edentulous patients. Clin Oral Implants Res. 2015 Oct;26(10):1121-8. doi: 10.1111/clr.12499. Epub 2014 Nov 5. PMID 25370914
- [Result] Bergenblock S, Andersson B, Furst B, Jemt T. Long-term follow-up of CeraOne single-implant restorations: an 18-year follow-up study based on a prospective patient cohort. Clin Implant Dent Relat Res. 2012 Aug;14(4):471-9. doi: 10.1111/j.1708-8208.2010.00290.x. Epub 2010 Jun 25. PMID 20586784
- [Result] Albrektsson T, Dahlin C, Jemt T, Sennerby L, Turri A, Wennerberg A. Is marginal bone loss around oral implants the result of a provoked foreign body reaction? Clin Implant Dent Relat Res. 2014 Apr;16(2):155-65. doi: 10.1111/cid.12142. Epub 2013 Sep 4. PMID 24004092